CLINICAL TRIAL: NCT00993902
Title: Double and Single Intrauterine Insemination In Controlled Ovarian Stimulation (COH) Cycles With Multifollicular Development
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Associated Prof.Tayfun Bagis, MD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BU1
Record Dates: First submitted 2009-07-22; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Infertility
Keywords: Double IUI; Intrauterine insemination; Unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single IUI (Sham Comparator): Single IUI will be carried on after 36-38 hours of HCG administration
  Interventions: Procedure: Intrauterine insemination (single)
- Double IUI (Active Comparator)
  Interventions: Procedure: Double intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination (single) — Single IUI after 36-38 hours of HCG
  Other Names: Group I
  Arms: Single IUI
Procedure: Double intrauterine insemination — Double insemination after 18 and 40 hours of HCG administration.
  Other Names: Grup II
  Arms: Double IUI

SUMMARY:
Our hypothesis is double insemination will improve pregnancy rates in coh cycles with more than one dominant follicles (>16mm).

DETAILED DESCRIPTION:
Metaanalysis for the effects of double IUI demonstrates that effects of this procedure is not different from single IUI. It is known that nearly 25% of coh cycles is evident by monofollicular development.For this reason it is possible that this monofollicular cycles in the studies could decrease the effects of double IUI.

Inclusion criteria:

1. Patients with unexplained infertility or mild male factor infertility whom admitted to the COH+IUI programme in our infertility unit.
2. Female age <37 years old.
3. Baseline FSH <12 mIU/L
4. Total antral follicle count>6
5. During the first three cycles of COH+IUI
6. Minimum 2 follicles >16 mm at the day of HCG.

Primary outcome:

Ongoing pregnancy rates

Secondary outcomes:

The effects of different coh regimens (CC,FSH,CC+FSH)on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained and mild male factor infertile patients
* Minimum 2 follicles >16 mm at the day of HCG
* First 3 cycles

Exclusion Criteria:

* Basal FSH >12 mIU/L
* Total antral follicle count<6
* Severe male factor infertility

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rates | pregnancy >12 weeks of gestation

SECONDARY OUTCOMES:
The effects of different coh regimens on outcomes | 14 days after IUI procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Medical Faculty Obstetric and Gynecelogy Department, Infertility and IVF unit, Adana, Turkey (Türkiye)

REFERENCES:
- [Derived] Bagis T, Haydardedeoglu B, Kilicdag EB, Cok T, Simsek E, Parlakgumus AH. Single versus double intrauterine insemination in multi-follicular ovarian hyperstimulation cycles: a randomized trial. Hum Reprod. 2010 Jul;25(7):1684-90. doi: 10.1093/humrep/deq112. Epub 2010 May 10. PMID 20457669